CLINICAL TRIAL: NCT03549689
Title: Effect of Reducing Nucleotide Exposure on Bone Health (ReNew)
Acronym: ReNew
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn by drug manufacturer
Sponsor: Philip Grant (Other)
Responsible Party: Sponsor-Investigator, Philip Grant, Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43453
Record Dates: First submitted 2018-04-26; First posted 2018-06-08 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: HIV/AIDS; HIV-1-infection; Osteopenia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Bone Diseases, Metabolic | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Switch (Experimental): Dolutegravir (DTG) 50MG/ lamivuidne (3TC) 300MG FIXED_DOSE COMBINATION (FDC) DAILY at randomization for 96 weeks
  Interventions: Drug: Dolutegravir (DTG) 50MG/lamivudine (3TC) 300MG FIXED DOSE COMBINATION (FDC)
- Continuation (Active Comparator): Continue current tenofovir alafenamide (TAF)-containing ART regimen from weeks 0 to 96.
  Interventions: Drug: Current tenofovir alafenamide (TAF)-containing ART regimen

INTERVENTIONS:
Drug: Dolutegravir (DTG) 50MG/lamivudine (3TC) 300MG FIXED DOSE COMBINATION (FDC) — Participants randomized to the Switch Arm will take DTG 50mg/3TC 300mg FDC once daily with or without food at approximately the same time each day.
  Arms: Switch
Drug: Current tenofovir alafenamide (TAF)-containing ART regimen — Continuation of current TAF-containing ART for 96 weeks.
  Arms: Continuation

SUMMARY:
This is an open-label, randomized pilot study to assess the effect on bone mineral density (BMD) of a switch from a tenofovir alafenamide-containing antiretroviral regimen to dolutegravir/lamivudine vs. a continuation of the tenofovir alafenamide-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by a positive 4th generation assay or by any licensed ELISA test kit confirmed by Western blot at any time prior to study entry.
2. Age ≥18 years
3. HIV-1 RNA BLQ (e.g., <20 copies/mL or other threshold based on the local viral load assay used) for at least 12 months prior to study entry excluding blips (i.e., a single measurement <200 copies/mL preceded and followed by measurements BLQ)
4. On a stable TAF-containing ART that also includes at least 2 other antiretrovirals, with no changes in the 12 months prior to entry (except for a switch to a co-formulated tablet from the component tablets or a switch from ritonavir to cobicistat)
5. Lumbar spine, femoral neck or total hip BMD T-score ≤-1.0 from a DXA scan within the past 48 weeks
6. If receiving testosterone or estrogen replacement therapy, on a stable dose for ≥3 months prior to enrollment without plan to change dose during the study period.
7. Acceptable blood laboratory values at screening visit:

   * CD4+ T-cell count ≥200 cells/µL
   * Phosphate ≥2mg/dL
   * 25-hydroxyvitamin D level ≥10 ng/ml
   * Calculated creatinine clearance (CrCl) ≥50 mL/min as estimated by the Cockcroft-Gault equation*:

     * For men = CrCl (mL/min) = (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dL x 72)

   For women, multiply the above result by 0.85
8. For women of reproductive potential, negative serum or urine pregnancy test prior to screening and a negative urine pregnancy test at the entry visit prior to randomization and agreeable to using a contraceptive of choice during the study period.

"Women of reproductive potential" are defined as women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months) and have not undergone surgical sterilization (i.e., hysterectomy, bilateral oophorectomy, or tubal ligation; participant report sufficient)

Exclusion Criteria:

1. Current systemic glucocorticoid use
2. Lumbar spine, femoral neck or total hip BMD T-score <-3.0
3. Previous, current pharmacologic treatment, or plan for initiation of therapy for osteoporosis (i.e., bisphosphonates, teriparatide, denosumab, tamoxifen or raloxifene)
4. Previous fragility fracture (i.e., any fall from a standing height or less that resulted in a fracture)
5. History of genotypic resistance or phenotypic resistance to either DTG or 3TC. The interpretation of genotypic resistance is based on output from the Stanford HIV Resistance Database (available at https://hivdb.stanford.edu). Isolates with an interpretation of low-level resistance or higher are considered resistant.
6. History of virologic failure (i.e., confirmed HIV-1 RNA level ≥200 copies/mL after over 6 months of therapy) while on an integrase inhibitor (i.e., raltegravir, elvitegravir, bictegravir, or dolutegravir) or on lamivudine/emtricitabine prior to study enrollment. Any antiretroviral history (even before routine virologic monitoring became standard of care) that would suggest the presence of the M184V mutation should be considered exclusionary
7. ALT ≥5 X ULN, OR ALT ≥3xULN and bilirubin ≥1.5xULN (with >35% direct bilirubin)
8. Severe hepatic impairment (Child Pugh Class C)
9. Anticipated need for antiviral therapy for HCV
10. Hepatitis B surface antigen positive or Hepatitis B DNA positive
11. Weight >300 pounds, precluding safe DXA testing
12. Breastfeeding, pregnancy, or plans to become pregnant during the study
13. Known allergy/sensitivity to DTG or 3TC.
14. Receipt or planned receipt of prohibited concomitant medications (See section 5.4)
15. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study procedures and treatment.
16. Any serious medical or psychiatric illness that, in the opinion of the site investigator, precludes safe participation or adherence to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in lumbar spine Bone Mineral Density (BMD) at 96 weeks | Baseline and 96 weeks
  Compare the percentage change from entry to 96 weeks in lumbar spine BMD in those randomized to DTG/3TC vs. those continuing a TAF-based regimen

SECONDARY OUTCOMES:
Percentage change in lumbar spine BMD at 48 weeks | Baseline and 48 weeks
  Compare the percentage change from entry to 48 weeks in lumbar spine BMD in those randomized to DTG/3TC vs. those continuing a TAF-based regimen
Percentage change in total hip BMD at 48 weeks | Baseline, 48 weeks
  Compare the percentage change from entry to 48 weeks in total hip BMD in those randomized to DTG/3TC vs. those continuing a TAF-based regimen
Percentage change in total hip BMD at 96 weeks | Baseline, 96 weeks
  Compare the percentage change from entry to 96 weeks in total hip BMD in those randomized to DTG/3TC vs. those continuing a TAF-based regimen
Change in CTX (a bone resorption marker) | Baseline, 12 weeks, 48 weeks, and 96 weeks
  Compare the changes in CTX from entry to 12, 48, and 96 weeks
Change in P1NP (a bone deposition marker) | Baseline, 12 weeks, 48 weeks, and 96 weeks
  Compare the changes in P1NP from entry to 12, 48, and 96 weeks
Change in urine β2-microglobulin (renal tubular marker) | Baseline, 48 weeks, and 96 weeks
  Compare the changes in urine β2-microglobulin from entry to 48 weeks and 96 weeks.
Change in urine RBP (renal tubular marker) | Baseline, 48 weeks, and 96 weeks
  Compare the changes in RBP from entry to 48 weeks and 96 weeks.
Change in urine protein | Baseline, 48 weeks, and 96 weeks
  Compare the changes in protein from entry to 48 weeks and 96 weeks.
Change in urine albumin | Baseline, 48 weeks, and 96 weeks
  Compare the changes in urine albumin from entry to 48 weeks and 96 weeks.
Change in fractional excretion in phosphate | Baseline, 48 weeks, and 96 weeks
  Compare the changes in fractional excretion of phosphate from entry to 48 weeks and 96 weeks.
Percentage change in total lean mass | Baseline, 48 weeks, and 96 weeks
  Compare the percentage change from entry to 48 weeks and 96 weeks in total lean mass (as measured by whole body DXA)
Percentage change in trunk fat | Baseline, 48 weeks, and 96 weeks
  Compare the percentage change from entry to 48 weeks and 96 weeks in trunk fat (as measured by whole body DXA)
Percentage change in limb fat | Baseline, 48 weeks, and 96 weeks
  Compare the percentage change from entry to 48 weeks and 96 weeks in limb fat (as measured by DXA)
Maintenance of HIV RNA level | 48 weeks and 96 weeks
  Compare the levels of HIV RNA <50 copies/mL and below the limit of quantification (BLQ) at 48 weeks and 96 weeks using the FDA snapshot algorithm
Grade 3 or 4 adverse events | 96 weeks
  Compare rates of grade 3 or 4 adverse events experienced by participants through 96 weeks
Treatment discontinuation of study medication due to adverse effect | 96 weeks
  Compare treatment discontinuation of study medication due to adverse effect experienced by participants through 96 weeks
Change in fasting lipids | Entry, 48 weeks, and 96 weeks
  Compare changes in fasting lipids (total cholesterol, LDL, HDL, and triglycerides) at entry, 48 weeks, and 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip Grant, MD, Principal Investigator — Stanford University
Locations (10):
- United States (10):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Emory, Atlanta, Georgia
  - Northwestern, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Columbia, New York, New York
  - Penn, Philadelphia, Pennsylvania
  - Dallas VA Medical Center, Dallas, Texas
  - UT Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided